CLINICAL TRIAL: NCT04768335
Title: Pilot Study: the Links Between Basic Auditory Processes and High Functioning Cognitive Processes in Schizophrenia (Reality Monitoring and Emotional Perception)
Brief Title: Auditory Processes and Emotional Perception in Schizophrenia
Acronym: AUDISPACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CSRM01
Record Dates: First submitted 2021-02-09; First posted 2021-02-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Basic Auditory Processes; Emotional Perception; Source Monitoring Deficits
Keywords: auditory processes; emotional perception; source monitoring; schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group with schizophrenia (Active Comparator): The schizophrenic subjects will undertake a 3 hour session of cognitive experiments. Tasks will include a battery of psychoacoustic tests, a source monitoring task, an externalization task, a pitch discrimination task and a speech-in-speech task.
  Interventions: Behavioral: cognitive experiments' session
- Healthy control subjects (Active Comparator): Healthy control subjects will undertake a 3 hour session of cognitive experiments. Tasks will include a battery of psychoacoustic tests, a source monitoring task, an externalization task, a pitch discrimination task and a speech-in-speech task.
  Interventions: Behavioral: cognitive experiments' session

INTERVENTIONS:
Behavioral: cognitive experiments' session — The aim of this unique session of cognitive experiments is to study the links between source memory deficits and externalization abilities in healthy control subjects. Results of this Arm 2 will be compared to those of Arm 1.

SUMMARY:
Schizophrenia is a mental illness with a variety of clinical symptoms that can be regrouped into 2 categories: positive and negative symptoms.

This mental illness is also characterised by cognitive alterations in various fields, including social cognition difficulties and self / non-self-discrimination difficulties.

Self and non-self-discrimination abilities have been regrouped under a function called source memory. This source memory enables a person to identify the source of an information previously encoded. In our everyday life, these processes are necessary to distinguish events generated by an external source from imagined events. It is called reality monitoring.

A number of studies have evidenced reality-monitoring alterations in patients suffering from schizophrenia. More specifically, patients would present with an externalisation bias, they would assign more imagined events to an external source. The knowledge of these deficits encourages the study of the processes involved in order to better understand the alterations, particularly including auditory processes. A recent study has shown that discrimination errors concerning certain sound characteristics (e.g. frequency) were associated to reality monitoring errors. However, the links between reality-monitoring and basic auditory processes have rarely been explored.

The dysfunction of the auditory "where" path, especially the possibility to discriminate between the intra and extra cephalic localisation of sounds, could lead to difficulties to discern between what is produced by one self and what is produced by another or the local environment.

DETAILED DESCRIPTION:
The main objective of this study is to study the links between source memory deficits and externalization abilities in schizophrenic patients and healthy subjects.

Also, this study will:

* evaluate the impact of emotional content on the ability to externalize an auditory perception
* evaluate the abilities to separate sources concerning vocal stimuli
* evaluate the basic auditory processes In order to meet the objectives, the correlation between the percentage of good attributions in the reality monitoring task and the percentage of correct perceptions in/out (sound perceived as coming from inside or outside the head) will be analyzed in the externalization task in patients suffering from schizophrenia.

Will also be analyzed:

* the number of correct perceptions In/Out in the externalization task
* the number of correct perceptions In/Out for the emotional stimuli
* the detection level of difference in pitch between 2 vocal sources pour the height discrimination task
* the number of correctly identified words in the speech-in-speech task

The tasks :

Subjects will undergo a battery of cognitive and auditory experiments in order to answer the objectives and hypothesis. The duration of the entire experiments will be 3.30 hours.

- Subjects will undergo the source monitoring task (30 min):

This task is divided in 2 parts:

* one part that will evaluate the reality monitoring performances (LISTENING task). Subjects either have to listen to words or imagine themselves listening to words
* another part evaluating internal source monitoring performances (SAY task). Subjects either have to pronounce words or imagine themselves pronouncing words.

  * In order to measure perception abilities, all subjects will undergo a battery of psychoacoustic tests (30 min) including the Tone Matching Task (TMT) which evaluates the capacity of discriminating static pitch. The battery is also composed of tasks measuring length, amplitude, etc…
  * A yes / no discrimination task will be used to measure the externalization abilities: subjects will have to discern whether a sound is perceived as coming from inside or outside the head
  * the ability to separate sources will be measured using 2 paradigms:
* a pitch discrimination task (30 min): it will evaluate the capacity to discern sources based on voice pitch
* a speech-in-speech task (30 min): target words are presented simultaneously to masks (composed of words time reversed so that have lost the semantic content). The subject has to listen and repeat the words heard.

ELIGIBILITY:
Inclusion Criteria:

Subjects aged between 18 and 65 years old - written given consent

For patients with schizophrenia:

- that meet the DSM-5.0 schizophrenia criteria

For healthy control subjects:

* absence of psychiatric disroders (past and actual) diagnosed according to the DSM-5.0
* absence of prodromal psychosis as measured by a score under 6 at the Prodromal Questionnaire PQ-16 (Ising et al., 2012)
* absence of auditory disorders (actual and past) (including tinnitus)
* absence of medical treatment (to the exception of contraceptive pills

Exclusion Criteria:

* history of neurological disorders or brain injury with loss of consciousness
* subjects presenting with highly developed musical abilities (frequently practicing a musical instrument)
* subjects presenting with an intellectual deficiency as measured by the Raven progressive matrices
* subjects under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Performance on a Reality monitoring task and on an externalization task | one day
  A computerized source memory task was designed for this study and a computerized externalization task was also designed (see description above). Rate of correct responses in both tasks is the main outcome.

SECONDARY OUTCOMES:
Performance on a task measuring the impact of emotional stimuli on externalization processes | one day
  computerized externalization task. Emotional nonverbal bursts are presented, the azimuth is varied in order to create the impression of the sound coming either from inside or outside the head. Subjects have to determine whether the emotional nonverbal burst was perceived as coming from inside or outside their head. The rate of correct responses (in / out) is the outcome.
Performance on source separating paradigms | one day
  2 computerized tasks.
  - Vocal pitch discrimination task (30 min): pairs of vocal vowels are presented, subjects will have to determine if the pairs differ in pitch or not.
  The rate of correct responses is the outcome.
  - Speech-in-speech task (30 min): target words are presented simultaneously to masks composed of time reversed words (having lost their semantic content). Subjects have to listen and repeat the words heard.
  The rate of correct words heard is the outcome.
Performance on basic auditory tasks | one day
  a computerized psychoacoustic battery of tests, including a Tone Matching Task (evaluating nonverbal pitch), and other psychoacoustic tasks measuring amplitude, length of sound etc… The rate of correct responses is the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No